CLINICAL TRIAL: NCT01093144
Title: Assessment of Pelvis Diameters as a Predictor for the Mode of Delivery ,Using Non-invasive, Ultrasound Based Measurements.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Trig Medical Inc (Industry)
Responsible Party: Tzipi Yakoby, Trig Medical Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP 006/2010
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Pregnancy; Women
Keywords: Delivery mode; pelvic measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: pelvic measurements using the LaborPro Device — pelvic measurements using the LaborPro Device,ultrasound non invasive measurements

SUMMARY:
Assessing the relation between the Pelvis diameters measured by the LaborPro, and the mode of delivery(normal vaginal delivery/instrumental delivery/Caesarean section.

DETAILED DESCRIPTION:
Assessing the relation between the Pelvis diameters measured by the LaborPro, and the mode of delivery(normal vaginal delivery/instrumental delivery/Caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* A subject is eligible to participate in the study if she meets all of the following inclusion criteria:
* Singleton pregnancy

  * Pregnant adult woman in labor
  * Willing to participate in the study and understands the study procedures

Exclusion Criteria:

* A subject is not eligible for participation in this study if he/she meets any of the following exclusion criteria scheduled for c/s active infection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
pelvis measurements influence on the Delivery mode | labor and delivery process
  pregnant woman's during a routine visit in the ultrasound unit will be requested to sign a concent and will undergo pelvic measurement using the LaborPro system.
  statistic analysis will ensue in order to ascertain the relationship between pelvic measurement and the mode of delivery.

SECONDARY OUTCOMES:
the influence of maternal parameters on delivery mode. | 1 year
  Assessing the influence of relevant obstetric and maternal parameters on delivery mode in relation to the study measured parameters

CONTACTS AND LOCATIONS:
Overall Officials: Yinon Gilboa, Dr, Principal Investigator — Tel Hashomer Medical Center
Locations (1):
- Shiba Medical Center, Tel Aviv, Israel